CLINICAL TRIAL: NCT04579692
Title: Phase 1 Clinical Trial for MR Guided Focused Ultrasound (FUS) Thalamotomy of Central Lateral Thalamic Nucleus for the Treatment of Medication-refractory Trigeminal Neuralgia
Brief Title: MR Guided Focused Ultrasound (FUS) for the Treatment of Trigeminal Neuralgia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Focused Ultrasound Foundation (Other); InSightec (Industry)
Responsible Party: Principal Investigator, Dheeraj Gandhi, Professor of Radiology, Neurology and Neurosurgery, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HP-00092927
Record Dates: First submitted 2020-09-28; First posted 2020-10-08 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Trigeminal Neuralgia
Keywords: Trigeminal pain; MR guided focused ultrasound
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- ExAblate Transcranial treatment (Experimental): The ExAblate Transcranial system will be used to destroy a small cluster of cells that may be causing the study participant's pain . The ExAblate uses ultrasound to heat a small spot in the brain called central lateral thalamic nucleus. Ultrasound passes through the skin and skull and into the brain to focus on this particular spot.
  Interventions: Device: ExAblate Transcranial treatment

INTERVENTIONS:
Device: ExAblate Transcranial treatment — Patients' head will be placed in ExAblate device to hold it still for the treatment. The ExAblate Transcranial helmet will be placed on their head. The investigators will measure the study participant's heart, blood pressure, temperature, and breathing rate before the treatment begins. MRI scans will be taken to make sure the ultrasound waves will be aimed exactly within the target. A series of MR images will be taken to identify the target area, and plan the study treatment. The study investigators will decide on the area of participant's brain that will be treated. The ExAblate Transcranial system will compute a plan to cover the treatment area. This area is gradually heated while monitoring the patient's responses and neurologic examination.
  Other Names: The ExAblate® MR guided focused ultrasound system

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of MRI-guided focused ultrasound (MRgFUS) for treating Trigeminal Neuralgia. Trigeminal Neuralgia (pain) is a type of pain involving the face that can be disabling to those it affects.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety and effectiveness of MRI-guided focused ultrasound (MRgFUS) for treating Trigeminal Neuralgia. Trigeminal Neuralgia (pain) is a type of pain involving the face that can be disabling to those it affects.

Usually, people with trigeminal pain receive medicines to control the pain. However, these medications may not give adequate pain relief. They may have unwanted side effects. In many patients with Trigeminal Neuralgia, a blood vessel compressing the nerve could be responsible for this condition. In such patients, surgery (also called micro-vascular decompression) is considered to be the best option if the medications do not control the pain. However, not all patients are good candidates for surgical correction and some patients may have recurrence of pain following surgical correction.

When surgery is not possible or recommended, other procedures are also available to patients. Such procedures usually result in selective damage to the nerve pain fibers in the Trigeminal nerve. Examples of these treatments include injection of materials such as Glycerol into the nerve, compression of the nerve with a balloon or selective radiation treatment of the nerve (stereotactic Radiosurgery). These treatments may not always improve the patient's pain or may only relieve the pain for a short duration of time.

These treatments may also result in damage to the nerve fibers that carry sensation from the face.

Our study will assess a new device for treating patients who have disabling pain that has not responded to medications or medications along with surgery. The device we will assess is called the ExAblate Transcranial focused ultrasound system. In this study, we will use this device to send ultrasound waves through the skull to precisely target and treat a tiny area of the brain called central lateral nucleus.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical Diagnosis of Classical or Idiopathic TN refractory to medical therapy
2. Age greater than 21 and less than 75 years
3. Subjects who are able and willing to give consent and able to attend all study visits
4. Documented chronic, severe pain for more than 6 months duration
5. Failure to respond to the usual therapeutic regimen considered to be standard of care for Trigeminal Neuralgia. The patient should have failed a trial of at least two classes of therapeutic agents, including an anticonvulsant agent
6. Patient with Trigeminal Neuralagia who has either failed a prior surgical approach considered to be standard of care for TN (Micro-vascular decompression, radiofrequency, stereotactic, Radiosurgery or glycerol) or is not considered to be an acceptable candidate for one of those alternative options (due to anesthesia risk, medical comorbidities or Patient refusal despite counseling).
7. Central lateral thalamotomy is feasible based on evaluation of imaging studies
8. Patient able to communicate sensations during the Exablate TcMRgFUS treatment
9. Two members of the medical team have agreed upon inclusion and exclusion criteria.

Exclusion Criteria:

* Patient with contra-indications to MRI such as severe claustrophobia and metallic implants incompatible with MRI.

  1. Severe psychiatric disorder such as uncontrolled depression, bipolar disorder, prior attempt at suicide or suicide ideation in preceding 12 months
  2. Life expectancy less than 12 months
  3. Anticoagulant or antiplatelet medications as well as underlying coagulopathy
  4. Prior or currently implanted thalamic DBS
  5. Pregnant ladies or women of childbearing age who are sexually active and not using contraception
  6. Inability to provide informed consent, for example due to underlying cognitive impairment or aphasia
  7. Presence of intracranial mass or an acute intracranial abnormality
  8. Subjects with unstable cardiac status such as Unstable angina pectoris, documented myocardial infarction within 6 months of protocol entry and ejection fraction less than 40
  9. Subjects exhibiting any behavior(s) consistent with ethanol or substance abuse as defined by the criteria outlined in the DSM-IV.
  10. Severe hypertension (diastolic BP > 100 on medication or persistently elevated SBP>140 mmHg despite adequate antihypertensive medications)
  11. History of immunocompromise including those who are HIV positive.
  12. History of intracranial hemorrhage, traumatic brain injury or thalamic stroke.
  13. Cerebrovascular disease (multiple CVA or CVA within 6 months)
  14. Subjects with life-threatening systemic disease that include and not limited to the following will be excluded from the study participation: HIV, Liver Failure, blood dyscrasias, etc.
  15. Subjects with a history of seizures within the past year
  16. Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment (can be up to 4 hours of total table time.)
  17. Are participating or have participated in another clinical trial in the last 30 days
  18. Skull Density Ratio (SDR) less than 0.4 ± 0.05
  19. History of multiple sclerosis.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment related adverse events | All events will be reported up to 6 months from treatment
  Procedure related or device related adverse events will be reported, from the treatment day through the 6-month follow-up period.

SECONDARY OUTCOMES:
Change in pain intensity | 6 months
  Efficacy of ExAblate TcMRgFUS for Thalamotomy will be evaluated using Barrow Neurological Institute (BNI) pain intensity score.
Change in pain intensity | 6 months
  Efficacy of ExAblate TcMRgFUS for Thalamotomy will be evaluated using Brief Pain Inventory-Facial.
Change in pain intensity | 6 months
  Efficacy of ExAblate TcMRgFUS for Thalamotomy will be evaluated using Pain Numeric rating scale (NRS).
Change in patient's perception of the effect of the procedure | 6 months
  Patient Global impression of change (PGIC): The effect of the procedure on patient perceived impact of pain related symptoms, emotions and quality of life will be measured using PGIC scale.

CONTACTS AND LOCATIONS:
Overall Officials: Dheeraj Gandhi, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No